CLINICAL TRIAL: NCT01504477
Title: A Phase I/II Clinical Trial of the Anti-EGFR Monoclonal Antibody, Panitumumab, and the Proteosomal Inhibitor, Bortezomib, in Patients With Advanced, Refractory KRAS Wild-Type Colorectal Cancer
Brief Title: Panitumumab and Bortezomib for Patients With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual--unable to meet accrual goals
Sponsor: Georgetown University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-033; X05374 (Other: Millennium Pharmaceuticals)
Record Dates: First submitted 2011-12-14; First posted 2012-01-05 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; relapsed; refractory; Kras wild type
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence | interventions — Panitumumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of Panitumumab and Bortezomib (Experimental): IV panitumumab and bortezomib
  Interventions: Drug: Panitumumab and bortezomib

INTERVENTIONS:
Drug: Panitumumab and bortezomib — Panitumumab 6 mg/kg IV over 60 minutes on Day -14 (first cycle only), then Day 1 and 15 of each 28-day cycle.
  Bortezomib will be administered in escalating doses until the maximum tolerated dose is determined and then at the maximum tolerated dose as an IV bolus injection over 3-5 seconds on Day 1, 8, and 15 of each 28-day cycle.
  Other Names: Velcade; Vectibix

SUMMARY:
Panitumumab plus bortezomib for colon cancer

DETAILED DESCRIPTION:
This study is for patients with colon cancer that cannot be fully removed by surgery and has come back after or not responded to standard chemotherapy treatment.

Subjects will be enrolled to either the first part of the study (Phase I) or the second part of the study (Phase II). Phase I will be completed before Phase II will start. The purpose of the Phase I part is to find the highest dose of bortezomib that can be given with panitumumab without causing severe side effects. The purpose of the Phase II part is to test the effects the two drugs have on subjects with colorectal cancer.

Panitumumab is a drug that targets a protein important for the growth of cancer cells known as EGFR. By blocking the activity of the protein, panitumumab can block cancer cell growth and even lead to their death. Panitumumab is given intravenously once every two weeks. Panitumumab is approved by the FDA for patients with colorectal cancer.

Bortezomib is a drug that targets a part of the cancer cell known as the proteosome. By inhibiting the proteosome, bortezomib can inhibit cancer cell growth and even lead to their death. Bortezomib is given intravenously, once a week, 3 out of every 4 weeks. Bortezomib is not FDA approved for the treatment of colorectal cancer.

As part of this study the investigators will be taking biopsies of patients' tumors before any treatment, after starting with the panitumumab alone, and after receiving both the panitumumab and bortezomib. The investigators want to investigate what markers inside tumors may relate to how well these two medications work. These biopsies are required as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal cancer with measurable or evaluable disease
* KRAS wild-type colorectal cancer
* Progression on, or intolerance of, or ineligibility for all standard therapies
* Progression on prior anti-EGFR therapy
* Lesion that is amenable to biopsy
* ECOG performance status 0-2
* LVEF >/= institutional normal
* Corrected QT interval less then 500 milliseconds by EKG
* Grade 2 or less peripheral neuropathy
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time must be </= 1.5 x upper limit of institution's normal range and INR < 1.5. Subjects on anticoagulants will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator.
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intracranial disease and have not had treatment with steroids within 1 week of study enrollment.
* Life expectancy > 12 weeks
* Subject is capable of understanding and complying with parameters of the protocol and able to sign and date the informed consent form.

Exclusion Criteria:

* CNS metastases which do not meet the criteria above
* Prior cancer chemotherapy, radiation therapy, or any investigational agent within three weeks before starting therapy
* Active severe infection or known chronic infection with HIV or hepatitis B virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
* Peripheral neuropathy >/= Grade 2 at baseline or peripheral neuropathy >/= Grade 1 with neuropathic pain
* Life-threatening visceral disease or other severe concurrent disease
* Female subject is pregnant or lactating
* Diagnosed or treated for another malignancy within 3 years of enrollment with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy
* Patient has hypersensitivity to bortezomib, boron, or mannitol
* Clinically significant and uncontrolled major medical condition(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan for this

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination of Panitumumab and Bortezomib: IV panitumumab and bortezomib
  Panitumumab and bortezomib: Panitumumab 6 mg/kg IV over 60 minutes on Day -14 (first cycle only), then Day 1 and 15 of each 28-day cycle.
  Bortezomib will be administered in escalating doses until the maximum tolerated dose is determined and then at the maximum tolerated dose as an IV bolus injection over 3-5 seconds on Day 1, 8, and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Combination of Panitumumab and Bortezomib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.83 (5.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose of bortezomib (to be used in combination with panitumumab)
Time Frame: 12 months
Population: The maximally tolerated dose of bortezomib weekly to be used in combination with with Panitumumab every 2 weeks
Measure: Number; unit: mg/m2
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
mg/m2 | 1.6

2. Secondary Outcome: Percent of Patients With Disease Control
Description: Stable disease after 2 cycles, partial response or complete response as determined by RECIST v1.0
Time Frame: 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
percentage of participants | 0

3. Secondary Outcome: Percent of of Patients With a Complete or Partial Response
Description: Partial response plus complete response as per RECIST v1.0
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Duration of Disease Control
Description: Time from study registration until progressive disease
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
Days | 35.5 [8 to 47]

5. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose of panitumumab (to be used in combination with bortezomib)
Time Frame: 12 months
Population: The maximum tolerated dose of panitumumab (to be used in combination with bortezomib)
Measure: Number; unit: mg/kg
Arm/Group | Combination of Panitumumab and Bortezomib
Number analyzed (Participants) | 6
mg/kg | 6

ADVERSE EVENTS:
Arm/Group | Combination of Panitumumab and Bortezomib
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Panitumumab and Bortezomib (N=6)
fatigue (General disorders) | 2 — CONSTITUTIONAL SYMPTOMS
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Electrolyte (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No